CLINICAL TRIAL: NCT00739661
Title: A Phase II, Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial Evaluating the Efficacy and Safety of Vismodegib (GDC-0449) As Maintenance Therapy in Patients With Ovarian Cancer in a Second or Third Complete Remission
Brief Title: A Study of Vismodegib (GDC-0449, Hedgehog Pathway Inhibitor) As Maintenance Therapy in Patients With Ovarian Cancer in a Second or Third Complete Remission
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHH4489g
Record Dates: First submitted 2008-08-21; First posted 2008-08-22 (Estimated); Results first posted 2012-04-26 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-05

CONDITIONS: Ovarian Cancer
Keywords: Systemic Hedgehog; Hedgehog Pathway Inhibitor
MeSH Terms: conditions — Ovarian Neoplasms | interventions — HhAntag691

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Vismodegib 150 mg (Experimental): Patients received vismodegib 150 mg orally once daily until radiographically confirmed disease progression, intolerable toxicity, or withdrawal from the study.
  Interventions: Drug: Vismodegib 150 mg
- Placebo to vismodegib (Placebo Comparator): Patients received placebo to vismodegib orally once daily until radiographically confirmed disease progression, intolerable toxicity, or withdrawal from the study.
  Interventions: Drug: Placebo to vismodegib

INTERVENTIONS:
Drug: Vismodegib 150 mg — Vismodegib 150 mg was provided in hard gelatin capsules.
  Other Names: GDC-0449
  Arms: Vismodegib 150 mg
Drug: Placebo to vismodegib — Placebo to vismodegib consisted of the excipients for vismodegib without the active molecule in hard gelatin capsules matching the active drug product in color and size.
  Arms: Placebo to vismodegib

SUMMARY:
The study was a Phase II, randomized, placebo-controlled, double-blind, multicenter clinical trial of vismodegib (GDC-0449) in patients with ovarian cancer in a second or third complete remission. Patients were randomized in a 1:1 ratio to either vismodegib or placebo. Randomization was stratified based on whether their cancer was in a second or third complete remission.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of epithelial ovarian carcinoma, primary peritoneal carcinoma, or fallopian tube carcinoma
* Must be in second or third complete remission, have received chemotherapy (platinum-based and/or non-platinum-based) for recurrent disease, and have achieved a complete remission after their most recent chemotherapy regimen. Complete remission is defined as no symptoms suggestive of persistent cancer, computed tomography (CT) scan of the chest/abdomen/pelvis without evidence of ovarian cancer within 4 weeks of randomization, and normal CA-125 (measured within 2 weeks of randomization) following completion of prior chemotherapy. The study investigator should confirm the status of disease remission by CT scan before patient enrollment. If patient has lymphadenopathy by CT scan and the investigator thinks that it is unlikely due to ovarian cancer, this patient is considered eligible. If indicated, a confirmatory biopsy should be performed.
* Patients must have completed their most recent cytotoxic chemotherapy regimen (platinum-based or non-platinum based) no less than 3 weeks and no more than 14 weeks prior to randomization.
* Archival tissue must be available and requested.
* Negative pregnancy test on Day 1 (first day the patient receives vismodegib or placebo).
* For women of childbearing potential: Use of two effective methods of contraception, including one barrier method.

Exclusion Criteria:

* Pregnancy or lactation.
* Patients whose ovarian cancer is in first remission.
* Patients must not have experienced more than two prior recurrences of disease.
* Concurrent non-protocol-specified anti-tumor therapy, either approved or unapproved (eg, chemotherapy, hormonal therapy, other targeted therapy, radiation therapy, surgery, herbal therapy). Hormonal replacement therapies for treatment of postmenopausal symptoms do not exclude patients from this study.
* Current, recent (within 4 weeks of Day 1), or planned participation in an experimental drug study while enrolled in this study.
* History of other malignancies within 3 years of Day 1, except for tumors with a negligible risk for metastasis or death, such as adequately treated basal cell carcinoma (BCC) or squamous-cell carcinoma of the skin; ductal carcinoma in situ of the breast; or carcinoma in situ of the cervix.
* Uncontrolled medical illnesses such as infection requiring intravenous (IV) antibiotics.
* Life expectancy < 12 weeks.
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or that might affect interpretation of the results of the study or render the patient at high risk from treatment complications.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2008-12 (Actual); Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josina Reddy, M.D., Ph.D., Study Director — Genentech, Inc.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vismodegib 150 mg | Placebo to Vismodegib
Started | 52 | 52
Completed | 6 | 10
Not Completed | 46 | 42
Not completed — Adverse Event | 2 | 0
Not completed — Physician decision to withdraw patient | 1 | 0
Not completed — Patient decision to withdraw | 9 | 4
Not completed — Disease progression, radiographic | 33 | 37
Not completed — Reason for discontinuation not available | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vismodegib 150 mg | Placebo to Vismodegib | Total
Number analyzed (Participants) | 52 | 52 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (10.2) | 58.6 (8.9) | 57.9 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 52 | 104
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time between randomization and disease progression, as confirmed by radiography, or death for any reason. Since patients were in remission at the start of the study, they had no evidence of the presence of tumors. Disease progression was defined as radiographic evidence of a tumor. Tumor assessments by computed tomography (CT) of the chest, abdomen, and pelvis were performed at screening and every 8 weeks during the study.
Time Frame: From randomization date through the data cut-off date of May 15, 2010, up to 100 weeks
Population: Intent-to-treat patient population: All randomized patients.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vismodegib 150 mg | Placebo to Vismodegib
Number analyzed (Participants) | 52 | 52
Months | 7.5 [5.59 to 11.24] | 5.8 [4.14 to 7.49]

2. Secondary Outcome: Progression-free Survival (PFS) in Patients With Versus Without Hedgehog Antigen Tumor Expression
Description: Hedgehog antigen expression was measured with immunohistochemical methods in tumor tissue taken from each patient prior to enrollment in the study. The percentage of cells with (> 0%) and without (0%) Hedgehog antigen expression was measured microscopically. PFS was defined as the time between randomization and disease progression, as confirmed by radiography, or death for any reason. Tumor assessments by computed tomography (CT) of the chest, abdomen, and pelvis were performed at screening and every 8 weeks during the study.
Time Frame: From randomization date through the data cut-off date of May 15, 2010, up to 100 weeks
Population: Intent-to-treat patient population: All randomized patients. Tissue for evaluation was only available for 29 patients in the vismodegib group and 28 patients in the placebo group.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vismodegib 150 mg | Placebo to Vismodegib
Number analyzed (Participants) | 29 | 28
Months
  0% of cells with hedgehog punctate stain | 7.00 (3.48) [3.48 to 8.05] | 5.32 [1.94 to NA] — The upper limit of the confidence interval could not be estimated due to the small sample size.
  > 0% of cells with Hedgehog punctate stain | 9.13 [1.81 to 11.24] | 7.36 [3.12 to 10.97]

3. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from randomization until death by any cause.
Time Frame: From randomization date through the data cut-off date of May 15, 2010, up to 100 weeks
Population: Intent-to-treat patient population: All randomized patients.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Vismodegib 150 mg | Placebo to Vismodegib
Number analyzed (Participants) | 52 | 52
Months | NA (NA) — The data were not mature for analysis. Only 2 deaths in the vismodegib group were reported as of the 15 May 2010 data cutoff. | NA (NA) — The data were not mature for analysis. Only 1 death in the placebo group was reported as of the 15 May 2010 data cutoff.

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were recorded starting at randomization until 45 days after the last dose of treatment or after the initiation of new anti-tumor therapy, whichever was earlier, up to 100 weeks.
Description: Adverse events were reported for the safety-evaluable population, which was defined as all patients who received at least one dose of study treatment.
Arm/Group | Vismodegib 150 mg | Placebo to Vismodegib
Serious Adverse Events (participants affected / at risk) | 6/52 | 3/52
Other Adverse Events (participants affected / at risk) | 51/52 | 44/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vismodegib 150 mg (N=52) | Placebo to Vismodegib (N=52)
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Chest Pain (General disorders) | 1 | 0
Device Related Infection (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1
Hepatic Enzyme Increased (Investigations) | 1 | 0
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal Colic (Renal and urinary disorders) | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vismodegib 150 mg (N=52) | Placebo to Vismodegib (N=52)
Nausea (Gastrointestinal disorders) | 17 | 9
Abdominal Pain (Gastrointestinal disorders) | 10 | 7
Constipation (Gastrointestinal disorders) | 12 | 5
Diarrhoea (Gastrointestinal disorders) | 6 | 8
Vomiting (Gastrointestinal disorders) | 8 | 5
Abdominal Pain Upper (Gastrointestinal disorders) | 9 | 3
Abdominal Discomfort (Gastrointestinal disorders) | 2 | 4
Abdominal Distension (Gastrointestinal disorders) | 2 | 4
Dry Mouth (Gastrointestinal disorders) | 5 | 1
Flatulence (Gastrointestinal disorders) | 2 | 4
Dyspepsia (Gastrointestinal disorders) | 3 | 2
Abdominal Pain Lower (Gastrointestinal disorders) | 3 | 1
Fatigue (General disorders) | 14 | 15
Asthenia (General disorders) | 5 | 3
Influenza (Infections and infestations) | 4 | 3
Urinary Tract Infection (Infections and infestations) | 3 | 0
Weight Decreased (Investigations) | 6 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 10 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 35 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 8
Back Pain (Musculoskeletal and connective tissue disorders) | 6 | 4
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 5 | 3
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 4 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2
Dysgeusia (Nervous system disorders) | 35 | 9
Headache (Nervous system disorders) | 5 | 6
Dizziness (Nervous system disorders) | 4 | 5
Neuropathy Peripheral (Nervous system disorders) | 2 | 4
Paraesthesia (Nervous system disorders) | 3 | 3
Ageusia (Nervous system disorders) | 4 | 1
Insomnia (Psychiatric disorders) | 3 | 3
Anxiety (Psychiatric disorders) | 3 | 2
Depression (Psychiatric disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 28 | 4
Rash (Skin and subcutaneous tissue disorders) | 6 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 3
Nail Disorder (Skin and subcutaneous tissue disorders) | 0 | 3
Hypertension (Vascular disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.